CLINICAL TRIAL: NCT04966546
Title: Targeting Spreading Depolarization After Chronic Subdural Hematoma Surgery (TASD)
Acronym: TASD
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Loss of Departmental support
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Andrew Phillip Carlson, Assistant Professor of Neurosurgery, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20-655
Record Dates: First submitted 2021-04-02; First posted 2021-07-19 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Chronic Subdural Hematoma
MeSH Terms: conditions — Hematoma, Subdural, Chronic | interventions — Memantine

STUDY DESIGN:
Intervention Model Description: Pilot parallel RCT
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only research pharmacist is unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Memantine (Experimental): Subjects will be given memantine 10mg PO/ NG BID for 7 days
  Interventions: Drug: Memantine Hydrochloride
- Placebo (Placebo Comparator): Subjects will be given identical placebo syrup PO/NG BID for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Memantine Hydrochloride — Active drug arm
  Arms: Memantine
Drug: Placebo — Simple syrup with peppermint oil added to match the commercial solution and make it indistinguishable
  Arms: Placebo

SUMMARY:
Chronic Subdural Hematoma (cSDH) is an extremely common problem, particularly in the aging population, where fluid like collections compress the brain, frequently requiring surgical drainage. After drainage, 25-50% of patients experience post operative neurologic deficits such as weakness or confusion that are often not explained by problems such as seizure, stroke, or mass effect from the fluid and blood. Recent subdural recordings have demonstrated that some of these neurological deficits may be related to waves of spreading depolarization (SD), which cause temporary neurological dysfunction. Our overall objective is to examine the relationship between neurological deficits and SD and to assess feasibility of a pilot trial to determine if a strategy of NMDA-R antagonism can effectively reduce SD and improve clinical recovery.

DETAILED DESCRIPTION:
1. Objectives 1.1. Assess risk factors for SD and seizures 1.2. Compare clinical outcomes between patients with SD and without 1.3. Obtain preliminary data on safety and efficacy of Memantine in subjects with SD 1.4. Assess early temporal relationship between SD and neurological deficits 1.5. Compare clinical outcomes between subjects with seizure and without
2. Background

   Chronic subdural hematoma (cSDH) represents a unique phenotype of traumatic brain injury (TBI) occurring almost exclusively in elderly patients. Chronic Subdural Hematoma (cSDH) is estimated to become the most common condition treated by neurosurgeons by 2030(1). Surgical evacuation is the mainstay of treatment, and though most patients recover with a straightforward course, up to 50% of patients develop postoperative neurological deficits or impaired recovery (2, 3). Though some of these events may be related to seizures or other metabolic changes(3), we recently demonstrated that spreading depolarization (SD) is definitively demonstrated in at least 15% of patients after surgical evacuation and are closely linked to postoperative neurological deficits(4). NMDA-R antagonists are a promising treatment for inhibiting SD, and we performed the first prospective study demonstrating dose dependent inhibition of SD with ketamine(5). Further, a recent randomized controlled trial demonstrated efficacy of memantine (a related NMDA-R antagonist) in neurologic recovery after moderate traumatic brain injury (6). What is not known is whether postoperative neurologic deficits and subsequent impaired recovery are explained by an SD dependent mechanism. There is a critical need to assess this mechanistic link with SD and neurological recovery after cSDH evacuation in order to develop effective targeted therapies.

   Our long-term goal is to develop effective SD targeted therapies to improve recovery after cSDH evacuation and other neurologic injuries. The overall objective of this project, which is the necessary next step toward attainment of this long-term goal, is to assess for the overall relationship between SD and clinical outcomes. The central hypothesis is that SD plays a causal role in postoperative neurologic deficits after cSDH evacuation and therefore could be a therapeutic target. This hypothesis was formulated based on several key pieces of preliminary data: 1) We have demonstrated that SD occurs after cSDH evacuation and is closely related to postoperative neurological deficits. 2) We have demonstrated prospectively that a strategy of NMDA-R antagonism can inhibit SD after brain injury. The rationale that underlies the proposed research is that the temporal and long-term clinical outcomes, as they relate to SD, must be better defined. Further, in order to ultimately perform a randomized trial for efficacy, pilot data are needed to assess feasibility and appropriate outcome measures and timing.
3. Study Design 3.1. Observational study with nested randomized controlled trial 3.1.1. All subjects undergoing surgery for chronic or subacute subdural hematoma will be screened for participation. The determination of the nature of the Subdural Hematoma will be based on the characteristic radiographic CT appearance of hypo or iso-attenuation of fluid in the subdural space with or without membranes and with or without <50% acute component. A 1x6 recording electrode will be placed for clinical monitoring at the time of surgery and left in place for 1-2 days after surgery. This will allow for recording of spreading depolarizations and seizures. Seizures will be treated as clinically indicated and provide additional potential benefit for these subjects. Subjects will initially be enrolled in an observational study focused on identifying risk factors for SD and poor outcomes. If SD is detected, subjects who consent will be randomized to a nested blinded pilot trial of the effect of a 7 day course of Memantine 10 mg compared to identical placebo on both ECoG (electrocorticography) and clinical outcomes. Patients may or may not undergo middle meningeal artery embolization per standard clinical recommendation. This will not be affected by participation in the study in any way.

3.1.2. Dose Selection Rationale Memantine usually start as 5 mg and titrate up to maximum dose of 20 mg per day. In this trial we will randomize to Memantine vs Placebo with dose of 10 mg BID without titration. The lack of titration is based on the requirement for acute action rather than chronic actions over a short interval. The study by Mokhtari et al used the same approach without titration. Multiple additional studies with similar and higher dose Memantine without titration are summarized in below table.

Published studies with higher dose Memantine without titration:

Study Design Population Indication Dose(s) Duration Adverse Events Mokhtari, 2018 RCT Moderate TBI Neurologic Recovery 30mg PO BID (no titration) 7 days None reported (BP, temp, 02sat, serum Na, Serum glu similar between groups) Bisaga, 2001 RCT Opioid depencance Opioid physical dependance 60mg PO prior to naloxone challenge Single dose None (BP, HR, 02 sat similar. Improved withdrawal symptoms after naloxone admin) Swerdlow, 2009 RCT Normal volunteers undergoing prepulse inhibition and startle testing n/a 20 or 30mg Single dose Dizziness at 30mg (no effect of drowsiness, queasiness, autonomic measures) Hart, 2002 RCT Healthy volunteers Discrimination of methamphatamine dosing 40mg Single dose None, less irritability with memantine Collins, 2007 RCT Cocaine users Cocaine pretreatment 60mg Single dose Increased "anxious" and "stimulated" reported effects during subsequent cocaine use Handforth, 2010 Single arm pilot trial Adults with tremor Tremor reduction Up to 40mg/day 16 wk Dizziness, HA, malaise, loss of consciousness, somnolence, weight gain, poor energy, imbalance, worse tremor Ferguson, 2007 Open label study with flexible dose Major depressive disorder Depressive symptoms Up to 40mg/day 10 weeks Somnolence, dizziness, insomnia Cekman, 2011 Case report Overdose Unintended 2000mg Single dose Sleepiness and coma. Tachycardia, hypertension, respiratory alkalosis, seizure.

Treated with plasmapheresis and DC home without sequelae

3.1.3. Allocation of Treatment and Randomization This is a nested Randomized Double Blinded Study within the observational study, once the SD is detected, subjects who consent will be randomized to a nested blinded pilot trial of the effect of a 7 day course of memantine 10 mg BID compared to identical placebo on both ECoG and clinical outcomes. The research pharmacist will be the only unblinded participant unless any safety concerns arise. All other study-related personnel, hospital care givers, and the patient will remain blinded.

ELIGIBILITY:
Inclusion Criteria:

* Surgical intervention for chronic or subacute SDH
* Electrode strip placed at time of surgery (for clinical indication of enhanced seizure monitoring)
* Age 18-100
* SD detected within 48h of surgery

Exclusion Criteria:

* Acute SDH requiring large craniotomy (some acute subacute component within cSDH is acceptable)
* Strip not feasible or safe to place at conclusion of surgery
* Known or suspected infection
* Recurrent surgery
* Subjects who previously participated in the study (contralateral or recurrent hematoma)
* Severe renal impairment (CrCl 5-29)
* Use of other NMDA antagonist
* Severe hepatic impairment
* Child-Pugh Class C hepatic impairment
* Known allergy to memantine
* Memantine use at time of admission
* Inability to obtain enteral feeding (oral or via NGT)
* Patients on acetylcholinesterase inhibitors
* Women of child-bearing age who are unwilling to undergo dual contraception for 30 days.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Spreading depolarizations and seizures | 5 days
  Neurophysiology: spreading depolarization rate, incidence, and duration before and after memantine and between groups.
90 day eGOS | 90 days
  "extended Glasgow outcome scale" 1-8 ordinal scale. * is the best.

SECONDARY OUTCOMES:
Neurological deficits: Incidence of new motor weakness or new dysphagia | 5 days
  Incidence of new motor weakness or new dysphagia during the first 5 post op days.
Safety | up to 90 days
  Incidence of treatment emergent adverse events, specifically dizziness, headache, confusion, and constipation, which have previously been associated with memantine.

CONTACTS AND LOCATIONS:
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: Undecided
We do not anticipate generating any unique resources during the completion of the aims of this proposal.
  The PI and team are strongly committed to the sharing of resources, experimental details and findings, in order to facilitate replication studies and collaboration. We will therefore make the results and procedures from our study widely available. This will include dissemination through the COSBID network of SD investigators (www.cosbid.org), presentations at national meetings focused on brain injury, and study results will be submitted for publication in peer-reviewed journals and made available via PubMed Central.